CLINICAL TRIAL: NCT01213602
Title: Bilateral Bispectral Index Changes During Knee Replacement Surgery With and Without Femoral Block
Brief Title: Bilateral Bispectral Index (BIS)-Monitoring in Trauma Surgery
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Hospital Universitari de Bellvitge, Anesthesiology Department
Other Study IDs: SAB-ANE-2010-01
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-02

CONDITIONS: Knee Replacement Surgery
Keywords: Trauma patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Femoral block preoperative: In one group (T1) with performance of femoral block before general anesthesia and administration of bolus of local anesthetic through stimulating catheter (combined anesthesia)
- Femoral block postoperative: In second group (T2) with a administration of local anesthetic through stimulating femoral catheter until awareness of patient (balanced anesthesia).

SUMMARY:
The principal objective is to notice the relevance of timing performance of femoral block for knee replacement surgery during general anesthesia and analyze the relationship with bilateral bispectral index (BIS) monitoring during induction and maintenance of anesthesia. Otherwise the investigators try to investigate if the timing of performance of this block influence in postoperative variables as pain or blood loss.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

ASA IV, patients with difficult airway management, patients with antecedent of cerebral ischemia, presence of atrioventricular fistula, patients with absent distal pulses or history of vascular surgery in the involved limbs, patients with high risk of deep vein thrombosis.-

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA physical status I-III patients scheduled for total knee arthoplasty
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Sevoflurane requirements | 6 months
  Combined ( femoral block and general anesthesia) or balanced anesthesia ( intravenous analgesics and general anesthesia) is evaluated on the requirements of inhalational hypnotics during surgery. Schedule time when BIS has to be in proper range (40-60): T1 T2 T3 T4 T5 T6
  T1 Induction T2 Inflated cuff ischemia T3 Incision T4 Unlocking cuff ischemia T5 End surgery T6 Time to wake the patient from the close of the sevoflurane vaporizer
  Each time include a period of adjustment in 5 minutes

SECONDARY OUTCOMES:
Intraoperative and postoperative opiates requirements and relations with CVI | Time surgery and 24,48 and 72 h postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Sabate Pes, MD PhD DEEA, Principal Investigator — Hospital Universitari Bellvitge
Locations (1):
- Antoni Sabate Pes, L'Hospitalet de Llobregat, Barcelona, Spain